CLINICAL TRIAL: NCT06460155
Title: CompuFlo CathCheck; Using Pulse Wave Analysis Versus the Epidurogram for Determining Epidural Catheter Location, A Crossover Study
Brief Title: CompuFlo CathCheck
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANES-2024-32648
Record Dates: First submitted 2024-05-07; First posted 2024-06-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Epidural Placement
Keywords: Epidural

STUDY DESIGN:
Intervention Model Description: This study is a prospective diagnostic accuracy study. All participants will undergo all three methods being studied: epidurogram (gold standard), CompuFlo CathCheck, and physical exam in PACU following epidural placement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Device: 3 methods intervention

INTERVENTIONS:
Device: 3 methods intervention — Stu All participants will undergo all three methods being studied: epidurogram (gold standard), CompuFlo CathCheck, and physical exam in PACU following epidural placement.

SUMMARY:
The purpose of this study is to determine if the Compuflo CathCheck system is equivalent to an epidurogram in determining epidural catheter location (in or outside the epidural space), using the epidurogram as the gold standard. In short, this will be completed by performing an epidurogram (as is standard of practice and the gold standard of determining epidural placement) and compare it to the results of the Compuflo CathCheck system. Equivalency will be summarized through agreement and concordance. Additionally, secondary outcomes will look at how classical physical exam findings to confirm epidural placement correlate and compare to epidurogram and Compuflo CathCheck findings.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patients (age 18-99 years old) undergoing epidural placement for an operative procedure will be eligible for participation in this study.

Exclusion Criteria:

* All patients unable to receive or who refuse placement of epidural will be excluded
* patients who are unable to consent
* non-English speakers, pregnant individuals)
* Individuals with known or who have an allergic reaction to bupivacaine

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CompuFlo's Success | baseline
  The measure is a binary outcome: the epidural catheter is in the epidural space or not.
  Each modality assessed will either conclude positive (in the correct space) no negative (notnint he correct space) There is no "value". The tools used for the assessment is actually what is being studied, compuflo, meniscus test, physical exam and epidurogram.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Berg, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States